CLINICAL TRIAL: NCT07245303
Title: Neural Mechanisms of Light Driven Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-2288; RM1NS140200-01 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain; Fibromyalgia; Healthy Controls Group - Age and Sex-matched
Keywords: functional connectivity; colored light analgesia; functional magnetic resonance imaging; quantitative sensory testing
MeSH Terms: conditions — Musculoskeletal Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Light stimuli will be presented in random sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Light Sequence 1 (Experimental): The sequence of stimulus presentation for resting state scans will be Static Green for 8 minutes then Equal Energy White for 8 minutes then S-cone modulating stimuli for 8 minutes.
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus
- Light Sequence 2 (Experimental): The sequence of stimulus presentation for resting state scans will be Equal Energy White for 8 minutes then Static Green for 8 minutes then S-cone modulating stimuli for 8 minutes.
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus
- Light sequence 3 (Experimental): The sequence of stimulus presentation for resting state scans will be Equal Energy White for 8 minutes then S-cone modulating for 8 minutes then Static Green stimuli for 8 minutes
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus
- Light Sequence 4 (Experimental): The sequence of stimulus presentation for resting state scans will be Equal Energy White for 8 minutes then S-cone modulating for 8 minutes then Static Green for 8 minutes
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus
- Light Sequence 5 (Experimental): The sequence of stimulus presentation for resting state scans will be S-cone modulating for 8 minutes then Static Green for 8 minutes then Equal Energy White stimuli for 8 minutes
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus
- Light Sequence 6 (Experimental): The sequence of stimulus presentation for resting state scans will be Static Green for 8 minutes, S-cone modulating for 8 minutes, then Equal Energy White for 8 minutes
  Interventions: Other: S-cone modulating visual stimulus; Other: Equal Energy White Visual Stimulus; Other: Green light visual stimulus (S-OFF); Other: Evoked Pressure Pain Stimulus

INTERVENTIONS:
Other: S-cone modulating visual stimulus — The investigators will deliver a uniform wide-field, S-cone modulating stimulus via a fiberoptic, MRI-safe visual stimulator. This stimulus approximates the appearance of white but modulates the S-cone, driving the S-ON and S-OFF pathways by alternating two lights at 19 Hz using a mixture of light emitting diodes (LEDs), including those embedded in our stimulus with spectral peaks of 405, 565, and 660 nm. This stimulus will differentially activate the S-cones where, between the two phases the ratio of S-cone activity is 100. The frequency alternating between the two lights, 19 Hz, was chosen because retinal ganglion cells in the retina still respond robustly but above the cortical perceptual flicker detection threshold.
Other: Equal Energy White Visual Stimulus — The investigators will deliver a uniform wide-field, equal-energy light stimulus via a fiberoptic, MRI-safe visual stimulator. This will serve as a reference condition in which chromatic opponency has been eliminated. This stimulus ensures that the quantal catch of each cone photoreceptor (S-, M- and L-) is held constant using a mixture of LEDs, including those embedded in our stimulus with spectral peaks of 405, 565, and 660 nm.
Other: Green light visual stimulus (S-OFF) — The investigators will deliver a uniform wide-field, green light modulating stimulus via a fiberoptic, MRI-safe visual stimulator. Static Green (565 nm) Light presented via MRI compatible light guides.
Other: Evoked Pressure Pain Stimulus — The pressure in which a rapid inflation cuff positioned over the left gastrocnemius achieves a pain severity of 40 where 0 is "no pain" and 100 is the "worst pain imaginable will be determined pre-scan and applied during the entire functional imaging acquisition to evoke a deep pressure pain.

SUMMARY:
The goal of this study will be to understand the biological mechanisms that are responsible to light-driven analgesia. Light presented to the retina has been shown to have pain relieving properties in pre-clinical and clinical studies. In this study the investigators will evaluate the functional connectivity between subcortical visual areas and non-image forming brain areas that are involved in pain sensation. The investigators will also evaluate how three colored light stimuli presented to the retina results in changes in whole brain evoked activation patterns in participants with chronic musculoskeletal pain and in healthy controls. The investigators will also assess while brain evoked activation patterns in response to a pressure pain stimulus in the presence of three light stimuli in individuals with chronic musculoskeletal pain and healthy controls.

DETAILED DESCRIPTION:
The investigators will recruit 30 participants with chronic musculoskeletal pain (cMSP) and 30 healthy, matched controls. Participants will undergo a comprehensive assessment of important covariates that influence pain experience. Individuals will then undergo quantitative sensory testing that will be used to psychophysically assess pain sensitivity and conditioned pain modulation (CPM) immediately prior to the scanning session. Individuals will then undergo fitting of a rapid inflation pressure cuff on the left calf to achieve the same level of pain among each participant (who may have different pain sensitivity). Once these settings are established, participants undergo MRI scanning per the protocol described below. Following each scan block, a brief pain assessment will be performed to determine pain severity (0-100 visual analog scale) to serve as a covariate for our proposed analyses (as pain can change over the course of imaging) and will enable correlation of BOLD signal change to pain in exploratory analyses designed to validate our mechanistic discoveries. The imaging data will then be pre-processed to ensure data quality and assurance and then analyzed to determine the functional connectivity and the evoked brain activation patterns.

ELIGIBILITY:
Inclusion Criteria for participants with cMSP and healthy controls (n=30)

* Adults ≥18 years of age.
* Individuals who do not have any plans for medication or treatment changes for the next 3 months.
* Participants must be willing and able to undergo an MRI.
* Participants must not be claustrophobic
* Participants must be alert and oriented and able to provide informed consent.
* Individuals must be able to speak and read English.

Inclusion Criteria for participants with cMSP only (n=30)

* To be eligible, participants must have a score of ≥7 on the Widespread pain index (WPI) and ≥5 on the symptom severity scale (SSS), or 4-6 on the WPI and ≥9 on the SSS in the 2016 Fibromyalgia Questionnaire.
* Pain symptoms must have been present for 3 months or longer.
* Pain must be present in 4 out of 5 body regions.
* Individuals enrolled will have an average pain severity ≥4 on the 0-10 NRS over the month prior to enrollment to recruit individuals with moderate to severe chronic MSP.

Inclusion Criteria for Participants with Congenital Stationary Night Blindness (n=2)

-2 additional participants without chronic MSP will be recruited with diagnosed congenital stationary night blindness

Exclusion Criteria:

* Presence of retinal vision disorders or conditions resulting in vision impairment.
* Patient-reported photosensitivity, photophobia, or aversion (as may occur in autoimmune diseases such as systematic lupus erythematosus).
* Disorders including uveitis, cataracts, color-blindness, history of seizure disorder.
* Plans for analgesic treatment plan changes in next 3 months (surgery, analgesic medication changes, injections, pain procedures, etc).
* Prisoner Status.
* Pregnancy.
* Contraindications to MRI imaging. These include the presence of implanted/embedded ferromagnetic materials, implanted medical devices that are not MRI compatible, and claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Resting State Functional Connectivity-seed Voxel Analysis in Participants with cMSP and Healthy Controls | During 8 minute resting state scan as part of the ~1 hour scanning session
  Functional connectivity assessed under three lighting conditions will be assessed with a seed voxel analysis with the seed region of interest set as the pregeniculate nucleus. A map of connectivity will be generated and displayed over inflated brain space. This map will be constructed by calculating the Fisher-transformed correlation coefficients between each voxel with the BOLD times series for the Pregeniculate nucleus. The higher the correlation coefficient, the stronger connectivity of each voxel to the pregeniculate. The correlation coefficient will be plotted as an map.
Whole Brain Evoked Activation Patterns in Response to Chromatic Stimuli Contrasted with Achromatic Stimuli in Participants with cMSP and Healthy Controls | During 6 minute functional imaging scan within the ~1 hour scanning protocol
  A generalized linear model (GLM) using Statistical Parametric Mapping (SPM) version 12 will be constructed. Blood oxygenation level dependent (BOLD) activation signal time series collected under the dynamic S-cone modulating stimulus condition will be contrasted to those collected during the equal energy stimulus condition. SPM will be used to create a contrast vector between the two conditions and a T-map will be created where the T-statistic for the contrast at each voxel will be plotted. The larger the t-statistic for each voxel the larger the contrast between the two light conditions.
Whole Brain Evoked Activation Patterns in Response to Chromatic Stimuli Contrasted with Achromatic Stimuli in Patients with cMSP and Healthy Controls Exposed to a Pressure Pain Stimulus | During 6 minute functional imaging scan within the 1 hour scanning protocol
  A generalized linear model (GLM) using Statistical Parametric Mapping (SPM) version 12 will be constructed. Blood oxygenation level dependent (BOLD) activation signal time series collected under the dynamic S-cone modulating stimulus condition will be contrasted to those collected during the equal energy stimulus condition in context of an evoked pressure pain stimulus. SPM will be used to create a contrast vector between the two conditions and a T-map will be created where the T-statistic for the contrast at each voxel will be plotted. The larger the t-statistic for each voxel the larger the contrast between the two light conditions.

SECONDARY OUTCOMES:
Pressure Pain Threshold | Within ~2 hours pre-scan
  Pressure Pain Threshold is the threshold in which pain is experienced in response to increasing force applied to the trapezius measured by a pressure algometer in kilograms of force per square centimeter (kgf/cm^2). The higher the value, the higher the threshold. The maximum is 10 kgf/cm^2 and minimum is 0.
Temporal Summation | Within ~2 hours pre-scan
  The investigators will evaluate temporal summation using a 40g Neuropen applied to the skin of the volar forearm and lumbar region, following a train of 10 identical stimuli (1 Hz). Participants will report retrospectively, the pain intensity of the 1st and 10th pinprick using a 0-10 numerical rating scale (NRS). 0 is the minimum and 10 is the maximum pain intensity that will be reported.
Conditioned Pain Modulation | Within ~2 hours pre-scan
  Conditioned Pain modulation magnitude will be calculated as the difference in mean pressure pain threshold (kgf/cm^2) measured prior to and during the conditioning stimulus (cold water bath), with increases in pressure pain threshold during conditioning interpreted as evidence of efficient endogenous pain inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mauck, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared at the time of manuscript publication at the end of the study within 1 year of completion. The data will be shared via the NIH HEAL Ecosystem. After the data is shared, there are no plans to stop sharing the data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the time of manuscript publication or within 1 year of study completion.
Access Criteria: The data will be made available on an NIH approved repository.